CLINICAL TRIAL: NCT06727305
Title: Characterization of mTOR Inhibitor Pharmacokinetics and Pharmacodynamics in Older Adults .
Brief Title: MTOR Inhibitors in Older Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Maryland, Baltimore (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Irina Timofte, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2024-0798; 1U01AG081450-01A1 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-12-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Aging; Geriatic; Disability
MeSH Terms: interventions — Sirolimus; Tablets; Everolimus

STUDY DESIGN:
Intervention Model Description: Patients who will be randomized in 1:1:1:1:1:1 ratios to receive oral tablet doses of sirolimus and everolimus with concentrations of 0.5mg, 1mg, 2mg each
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- sirolimus 0.5 mg Arm (Active Comparator): Participant would receive 0.5 mg of sirolimus.
  Interventions: Drug: Sirolimus 0.5 Mg Oral Tablet
- sirolimus 1 mg Arm (Active Comparator): Participant would receive 1 mg of sirolimus.
  Interventions: Drug: Sirolimus 1Mg Oral Tablet
- sirolimus 2 mg Arm (Active Comparator): Participant would receive 2 mg of sirolimus.
  Interventions: Drug: Sirolimus 2 MG Oral Tablet
- everolimus 0.5 mg Arm (Active Comparator): Participant would receive 0.5 mg of Everolimus.
  Interventions: Drug: Everolimus 0.5 MG Oral Tablet
- everolimus 1 mg Arm (Active Comparator): Participant would receive 1 mg of Everolimus.
  Interventions: Drug: Everolimus 1 MG Oral Tablet
- everolimus 2 mg Arm (Active Comparator): Participant would receive 2 mg of Everolimus.
  Interventions: Drug: Everolimus 2 MG Oral Tablet

INTERVENTIONS:
Drug: Sirolimus 0.5 Mg Oral Tablet — Sirolimus 0.5 mg oral tablets daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: sirolimus 0.5 mg Arm
Drug: Sirolimus 1Mg Oral Tablet — Sirolimus 1 mg oral tablets daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: sirolimus 1 mg Arm
Drug: Sirolimus 2 MG Oral Tablet — Sirolimus 2 mg oral tablets daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: sirolimus 2 mg Arm
Drug: Everolimus 0.5 MG Oral Tablet — Everolimus 0.5 mg oral tablets daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: everolimus 0.5 mg Arm
Drug: Everolimus 1 MG Oral Tablet — Everolimus 1 mg oral tablets daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: everolimus 1 mg Arm
Drug: Everolimus 2 MG Oral Tablet — Everolimus 2 mg oral tablets for daily for 2 weeks and complete PK/PD testing. After the first 2 weeks, dose increase, or dose reduction will be made to obtain a stable blood level of 5-7 ng/ml.
  Arms: everolimus 2 mg Arm

SUMMARY:
Over the past decades, healthcare systems face significant challenges to meet the needs of an aging population due to progressive debility, functional decline and chronic diseases development. While there is a growing appreciation of the potential impact of mTOR inhibitors on slowing aging processes, preventing chronic disease and prolonging healthy lifespan, a major challenge in developing clinical trials to establish the clinical efficacy of mTOR inhibitors is the absence of pharmacokinetics (PK) and pharmacodynamics (PD) data in older adults. The proposed study will provide the foundation for future clinical trials assessing the role of mTOR inhibitors on aging related indications

DETAILED DESCRIPTION:
Study Objectives To characterize Pharmacokinetics (PK) and Pharmacodynamics (PD) of mTOR Inhibitors and determine whether mTOR Inhibitors will improve phenotypic biomarkers of aging as measured by SASP (senescence-associated secretory phenotype) index score at 3 months follow-up in older adults.

Specific Aims:

Aim 1: To characterize Pharmacokinetics (PK) and Pharmacodynamics (PD) of mTOR Inhibitors (sirolimus and everolimus) in older adults.

Aim 2: To determine whether mTOR Inhibitors will improve phenotypic biomarkers of aging as measured by SASP (senescence-associated secretory phenotype) index score at 3 months follow-up.

Exploratory Aim 3: We will also assess the feasibility of collecting the laboratory biomarkers (ESR, CRP, S6K activity, mitochondrial function, metabolomics) and data regarding the functional biomarkers of aging measured by walking speed, chair stand, standing balance, grip strength

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling adults
2. Patients should be 65 Years and older
3. Patients is able to understand and follow trial procedures

Exclusion Criteria:

1. Creatinine clearance <30 mL/min;
2. History of chronic liver disease;
3. Uncontrolled Hypertension (i.e., systolic blood pressure >160 mm Hg);
4. Hemorrhagic central nervous system (CNS) event within 1 year from screening visit;
5. Thrombotic event (DVT,PE) within 1 year from screening visit if not on anticoagulation;
6. Planned major surgical procedures;
7. Cardiovascular diseases ( i.e., admission for heart failure or myocardial infarction within 12 months);
8. Taking medication that increase or decrease sirolimus blood concentrations;
9. Other investigational therapy received within 1 month prior to screening visit;
10. History of dementia; 11 Dependence in any Katz Basic Activities of Daily Living.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-11-13 (Estimated)

PRIMARY OUTCOMES:
Cmax for Sirolimus | Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24-hour post dose
  Maximum Sirolimus Concentration at Steady State (Cmax)
Cmax for Everolimus | Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 12-hour post dose
  Maximum Everolimus Concentration at Steady State (Cmax)
Ctrough for Sirolimus | Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24-hour post dose
  Trough Sirolimus Concentration at Steady State (Ctrough)
Ctrough for Everolimus | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 12-hour post dose
  Trough Everolimus Concentration at Steady State (Ctrough)
AUC for Sirolimus | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24-hour post dose
  Sirolimus Area Under the Curve from Time Zero to End of Dosing Interval (AUCtau) at Steady State
AUC for Everolimus | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 12-hour post dose
  Everolimus Area Under the Curve from Time Zero to End of Dosing Interval (AUCtau) at Steady State
CL/F for Sirolimus | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24-hour post dose
  Sirolimus Apparent Oral Clearance (CL/F)
CL/F for for Everolimus | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 12-hour post dose
  Everolimus Apparent Oral Clearance (CL/F)
S6K Activity, in Sirolimus cohorts | Predose (0 hour) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24-hour post dose on Day 1 and Day 14
  Pharmacodynamic parameter, S6K Activity, in Sirolimus cohorts
S6K Activity, in Everolimus cohorts | Predose (0 hour) on Day 14 and 0.5, 1, 1.5, 2.5, 3, 4, 6, and 12-hour post dose on Day 1 and Day 14
  Pharmacodynamic parameter, S6K Activity, in Everolimus cohorts
Senescence-associated secretory phenotype (SASP) index | Day 1 Week 1 (Baseline), Week 5, Week 9, Week 13
  Clinical biomarker parameter (SASP) index is a clinical biomarker parameter that measures the level of proteins secreted by senescent cells in the body.
Erythrocyte sedimentation rate (ESR) | Day 1 Week 1 (Baseline), Week 5, Week 9, Week 13
  Clinical biomarker parameter (ESR) is a blood test that detects and monitors inflammation in the body.
C-reactive protein (CRP) | Day 1 Week 1 (Baseline), Week 5, Week 9, Week 13
  A measure of Clinical biomarker parameter (CRP), is an inflammatory marker.
6-minute walk test (6MWT) | Day 1 Week 1 (Baseline), Week 5, Week 9, Week 13
  The 6MWT is simply a record of the distance (in meters) traveled by a given patient at his or her self-selected walking speed over a period of six minutes.
Short physical performance battery (SPPB) | Day 1 Week 1 (Baseline), Week 5, Week 9, Week 13
  Clinical biomarker parameter (SPPB) assesses lower extremity function in older adults. The test battery consists of three physical tasks (walking, sit-to-stand and balance) to assess functional mobility. The test will be performed according to standardized procedure. The maximal total score is 12 and higher total scores indicate a better lower extremity functioning.

SECONDARY OUTCOMES:
Change in SASP response at 3 months follow-up | Baseline, 3 months
  SASP (senescence-associated secretory phenotype) index score is quantified using blood work comparing results at baseline and at 3 months follow-up. Patients with high SASP scores have a poor survival rate, while patients with low SASP scores have a good survival rate.
Change in Laboratory Biomarker response (ESR) from baseline at 3 months follow-up | Baseline, 3 months
  Feasibility of collecting the laboratory biomarker - Erythrocyte sedimentation rate (ESR) is assessed by change in blood work readings ((millimeters per hour [mm/hour])) at 3 months follow-up.
Change in laboratory Biomarker response (CRP) from baseline at 3 months follow-up | Baseline, 3 months
  Feasibility of collecting the laboratory biomarker- C-Reactive Protein (CRP) is assessed by change in blood work readings (mg/dl) at 3 months follow-up.
Change in laboratory Biomarker response (S6K activity) from baseline at 3 months follow-up | Baseline, 3 months
  Feasibility of collecting the laboratory biomarker- S6 Kinase (S6K) activity is assessed by change in blood work readings (mg/dl) at 3 months follow-up.
Change in laboratory Biomarker response (mitochondrial function) from baseline at 3 months follow-up | Baseline, 3 months
  Feasibility of collecting the laboratory biomarker (mitochondrial function) is assessed by change in blood work readings at 3 months follow-up. The mitochondrial function will be measured through the Bioenergetic Health Index. The Bioenergetic Health Index (BHI) is calculated using the following formula: BHI=(ATP-linked×reserve capacity)/(proton leak×non-mitochondrial) - as described by Chacko et al. The expected range is 0-100.
Change in laboratory Biomarker response (metabolomics) from baseline at 3 months follow-up | Baseline, 3 months
  Feasibility of collecting the laboratory biomarker (metabolomics) is assessed by change in blood work readings at 3 months follow-up. Changes in blood metabolomics are quantified by measuring the concentration levels of individual metabolites within a blood sample using techniques like mass spectrometry (MS) or nuclear magnetic resonance (NMR) spectroscopy, where the relative abundance of each metabolite is compared between different samples, allowing for identification of changes in metabolic pathways based on variations in metabolite levels. The unit of measure is "concentration", usually expressed in micromolar (µM) or millimolar (mM), as it represents the quantity of a specific metabolite per unit volume of the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Timofte, MD, MS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No